CLINICAL TRIAL: NCT01329874
Title: Comparison of the Anesthetic Efficacy in Mandibular Molars With Acute Irreversible Pulpitis With Either Conventional Inferior Alveolar or Gow-gates Nerve Block Techniques Plus Buccal or Lingual Infiltration
Brief Title: Anesthetic Efficacy of Gow-Gates Versus Conventional Inferior Alveolar Nerve Block Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Research Manager of Mashhad University of Medical Sciences, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 89549
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-01

CONDITIONS: Anesthesia; Reaction; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gow gates ,conventional block injection (No Intervention): Patients will be selected from a group with acute irreversible pulpitis in mandibular molars. Half of the patients randomly selected for receiving gow gates block injection and half will receive traditional inferior block injection by 3.6 ml Lidocaine plus epinephrine.Teeth with no response to anesthetizing will be randomly divided into two group of either buccal or lingual infiltration.
  Interventions: Procedure: Type of block injection
- Buccal infiltration, Lingual infiltration (No Intervention)

INTERVENTIONS:
Procedure: Type of block injection — Patients will be selected from a group with acute irreversible pulpitis in mandibular molars. Half of the patients randomly selected for receiving gow gates block injection and half will receive traditional inferior block injection by 3.6 ml Lidocaine plus epinephrine.Teeth with no response to anesthetizing will be randomly divided into two group of either buccal or lingual infiltration.
  Other Names: Gow Gates technique; Conventional inferior block injection
  Arms: Gow gates ,conventional block injection

SUMMARY:
The purpose of this study is to determine whether Gow Gates block injection is more effective than conventional alveolar nerve block in anesthetising mandibular molars with acute pulpitis.

DETAILED DESCRIPTION:
Pain management and adequate anesthesia are of critical importance for the endodontist. Traditionally, mandibular teeth are anesthetized via inferior alveolar nerve block (IAN). However, this technique provides a marginal success rate of 19-56% in patients with irreversible pulpitis.Gow Gates technique introduced in 1973 for anesthetizing of mandibular molars with more accuracy, success and safety.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular molars with acute irreversible pulpitis

Exclusion Criteria:

* Unhealthy patients
* Patients who had taken pain killer less than 4 hours before appointment

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Number of participant who will have pain following Gow gates or traditional inferior alveolar nerve block | 6 months
  All participant asked to show their pain degree on VAS for evaluation the efficacy of two different block injections and two different infiltrations ( Buccal and lingual) as supplementary injections.

SECONDARY OUTCOMES:
Heart rate monitoring | before and after block injections (day 1)
  These records will be monitored by pulse oximeter device

CONTACTS AND LOCATIONS:
Overall Officials: Jamileh Ghoddusi, D.D.S,M.S.c, Principal Investigator — Dental Research Center, Faculty of Dentistry, Mashhad University of Medical Sciences
Locations (1):
- Dept of Endodontics, Faculty of Dentistry, Mashhad, Khorasan Razavi, Iran